CLINICAL TRIAL: NCT00449150
Title: Cetrorelix Pamoate Intermittent Intramuscular (IM) Dosage Regimens in Patients With Symptomatic BPH: a 1 Year Placebo-controlled Efficacy Study and Long-term Safety Assessment
Brief Title: Cetrorelix (CET) Pamoate Regimens in Patients With Symptomatic Benign Prostatic Hypertrophy (BPH)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial did not meet primary efficacy endpoint for double blind phase.
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z033
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2011-06

CONDITIONS: Benign Prostatic Hypertrophy
Keywords: Cetrorelix
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — cetrorelix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Group A: CET 78 mg + 78 mg (Experimental): Treatment course 1: Cetrorelix 78 mg + 78 mg
  * Week 0: 52 mg CET (2 injections)
  * Week 2: 26 mg CET (1 injection)
  Treatment course 2:
  * Week 26: 52 mg CET (2 injections)
  * Week 28: 26 mg CET(1 injection)
    4 days with treatment, Day 1 of each indicated week, 6 injections in total per patient.
  Interventions: Drug: Cetrorelix 78 mg + 78 mg
- Treatment Group B: CET 78 mg + 52 mg (Experimental): Treatment course 1: Cetrorelix 78 mg + 52 mg
  * Week 0: 52 mg CET (2 injections)
  * Week 2: 26 mg CET (1 injection)
  Treatment course 2:
  * Week 26: 52 mg CET (2 injections)
  * Week 28: Placebo (1 injection)
    4 days with treatment, Day 1 of each indicated week, 6 injections in total per patient.
  Interventions: Drug: Cetrorelix 78 mg + 52 mg; Drug: Placebo
- Treatment Group C: Placebo (Placebo Comparator): Treatment course 1:
  * Week 0: placebo (2 injections)
  * Week 2: placebo (1 injection)
  Treatment course 2:
  * Week 26: placebo (2 injections)
  * Week 28: placebo (1 injection)
    4 days with treatment, Day 1 of each indicated week, 6 injections in total per patient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cetrorelix 78 mg + 78 mg
  Other Names: CET; AEZS-102
  Arms: Treatment Group A: CET 78 mg + 78 mg
Drug: Cetrorelix 78 mg + 52 mg
  Other Names: CET; AEZS-102
  Arms: Treatment Group B: CET 78 mg + 52 mg
Drug: Placebo
  Other Names: Placebo (PLA)
  Arms: Treatment Group B: CET 78 mg + 52 mg; Treatment Group C: Placebo

SUMMARY:
Benign Prostatic Hypertrophy (BPH) is a common and bothersome condition of aging men. It is characterized by an enlargement of the prostate occurring in human male over the age of 50 which increases in prevalence with age, and among those aged 50 to 80, about 40% report moderate or severe urinary symptoms of prostatism. The aim of treatment is to improve patients' quality of life which primarily depends on the severity of the symptoms of BPH. Current treatments of BPH have a benefit / risk ratio which leaves room for improvement.

For this study, study medication (Cetrorelix pamoate or placebo) is administered by injection in the buttocks (Intramuscular). All patients completing the double-blind portion (Week 0 to 52) are eligible to receive the active drug during the open-label part of the study (Week 52 to 90).

DETAILED DESCRIPTION:
The objectives of the study are to develop a safe and tolerable intermittent dosage regimen of cetrorelix pamoate that provides prolonged improvement in BPH-related signs and symptoms.

Patients will enter a 4-week run-in no-treatment observation period to confirm severity and stability of voiding symptoms based on the International Prostate Symptom Score (IPSS).

Patients will then be allocated to study drug in a double-blind, randomized, double-dummy, placebo-controlled fashion.

Patients will be administered an IM injection of study drug at Week 0, 2, 26 and 28 and will be followed up to Week 52.

Then, in an open label fashion, patients will be administered an IM injection of study drug at Week 52, 54, 78 and 80 and will be followed up to Week 90.

ELIGIBILITY:
Inclusion Criteria:

* Benign Prostatic Hyperplasia, based on medical history
* Voiding symptoms

Exclusion Criteria:

* Urgent need for prostate surgery or prior surgical treatment of the prostate or bladder
* Major organ dysfunction
* Eczema (atopic dermatitis) treated during the last 6 months
* Current or recent treatment with sexual hormone drugs or 5 α reductase inhibitors or botulinum toxin type a (Botox) within the last 6 months prior randomization or with α blockers or saw palmetto within the last 6 weeks prior to randomization
* Urologic disorders including neurogenic bladder dysfunction due to diabetes mellitus or documented neurologic disorder, urethral stricture disease or history of pelvic radiation therapy
* History of acute obstructive, infectious, or neurological disorders of the genitourinary tract within the last 3 months

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hebert Lepor, MD, Principal Investigator — NYU Langone Health
Locations (68):
- United States (46):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Urology Group of Westrn Arkansas, Fort Smith, Arkansas
  - South Orange County Medical Research Center, Laguna Hills, California
  - California Professionnal Research, Newport Beach, California
  - William G. Moseley, San Diego, California
  - West Coast Clinical Research, Tarzana, California
  - Western Clinical Research, Inc., Torrance, California
  - Urology Research Options, Aurora, Colorado
  - Urologic Oncology, Aurora, Colorado
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Connecticut Clincal Research Center, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Tampa Bay Medical Research, Clearwater, Florida
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Miami VACM, Miami, Florida
  - Florida Healthcare Research, Ocala, Florida
  - Florida Urologist Specialists, Sarasota, Florida
  - Southeastern Research Group, Tallahassee, Florida
  - Southwestern Medical Research Institute, Columbus, Georgia
  - Northwestern University Feinberg School of Medecine, Chicago, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Northeast Indiana Research, LLC, Fort Wayne, Indiana
  - Kansas City Urology Care, Overland Park, Kansas
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Myron I. Murdock M.D. LLC, Greenbelt, Maryland
  - Michigan Institute of Urology, Saint Clair Shores, Michigan
  - Washington University, St Louis, Missouri
  - Metropolitan Urological Specialists, St Louis, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Delaware Valley Urology, LLC, Woodlane, New Jersey
  - Urology Group Of New Mexico, Albuquerque, New Mexico
  - Medical & Clinical Research Associates, Bay Shore, New York
  - Urological Surgeons of Long Island, Clinical Research Division, Garden City, New York
  - New York University School of Medecine, New York, New York
  - University Urology, New York, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Northeast Urology Research, Concord, North Carolina
  - Parkhurst Research Oganization Inc., Bethany, Oklahoma
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Vanderbilt University medical Center, Nashville, Tennessee
  - Corpus Christi Urology Group, Corpus Christi, Texas
  - Urology Clinics of North Texas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Department of Urology, Dallas, Texas
  - Institute and the Texas Prostate Center, Houston, Texas
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Integrity Medical Research, Mountlake Terrace, Washington
- National Oncological Hospital, Sofia, Bulgaria
- Canada (14):
  - Southern Interior Medical Research Inc., Kelowna, British Columbia
  - Andreou Research Inc., Surrey, British Columbia
  - Can-Med Clinical Reserach Inc., Victoria, British Columbia
  - The Male / FemaleHealth and Research Center, Barrie, Ontario
  - Centre for Advanced Urological Research, Kingston, Ontario
  - Urologic Associates, Urologic Medical Research, Kitchener, Ontario
  - Canada Place Building, North Bay, Ontario
  - The Fe/Male Health Centers, Oakville, Ontario
  - University Health Network Princess Margaret Hospital, Toronto, Ontario
  - The Male Health Center, Toronto, Ontario
  - Urology South Shore Research, Greenfield Park, Quebec
  - CHUM, Hopital St-Luc, Montreal, Quebec
  - Dynamik Research, Pointe-Claire, Quebec
  - CRCEO, Québec, Quebec
- Germany (7):
  - ClinPharm International GmbH Prufzentrum Berlin, Berlin
  - ClinPharm International GmbH Prufzentrum Bochum, Bochum
  - ClinPharm International GmbH Prufzentrum Dresden, Dresden
  - ClinPharm International GmbH Prufzentrum Frankfurt, Frankfurt
  - ClinPharm International GmbH Prufzentrum Gorlitz, Görlitz
  - ClinPharm International GmbH Prufzentrum Leipzig, Leipzig
  - ClinPharm International GmbH Prufzentrum Magdeburg, Magdeburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetrorelix 78+78: 78+78 means 78 mg combining Week 0 (52 mg) and Week 2 (26 mg) + 78 mg combining Week 26 (52 mg) and Week 28 (26 mg)
- Cetrorelix 78+52: 78+52 means 78 mg combining Week 0 (52 mg) and Week 2 (26 mg) + 52 mg combining Week 26 (52 mg) and Week 28 (0 mg)
- Placebo: Placebo on Week 0, 2 26 and 28
Period: Overall Study
Arm/Group | Cetrorelix 78+78 | Cetrorelix 78+52 | Placebo
Started | 219 | 230 | 218
Completed | 173 (Subjects could have more than one reason for not completing.) | 177 (Subjects could have more than one reason for not completing.) | 171 (Subjects could have more than one reason for not completing.)
Not Completed | 46 | 53 | 47
Not completed — Adverse Event | 11 | 18 | 9
Not completed — Lack of Efficacy | 1 | 2 | 2
Not completed — Other | 16 | 13 | 14
Not completed — Withdrawal by Subject | 17 | 18 | 21
Not completed — Protocol Violation | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetrorelix 78+78 | Cetrorelix 78+52 | Placebo | Total
Number analyzed (Participants) | 219 | 230 | 218 | 667
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 109 | 126 | 111 | 346
  >=65 years | 110 | 104 | 107 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.86 (8.27) | 64.04 (7.54) | 64.20 (7.76) | 64.03 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 219 | 230 | 218 | 667
Region of Enrollment [Number; unit: participants]
  United States | 142 | 148 | 140 | 430
  Canada | 38 | 42 | 39 | 119
  Bulgaria | 11 | 12 | 12 | 35
  Germany | 28 | 28 | 27 | 83

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptoms Score (IPSS)
Description: The International Prostate Symptoms Score (IPSS) score of benign prostata hyperplasia (BPH) symptoms is calculated based on a patient questionnaire assessing 7 items (incomplete voiding, frequency, intermittency, urgency, weak stream, hesitancy, nocturia) on a scale from 0 (best) to 5 (worst); total range: 0 points (best) to 35 points (worst)
Time Frame: Baseline and 52 weeks
Population: The Intent-to-treat (ITT) population included all participants for whom at least one post-baseline efficacy assessment was available; imputation per Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cetrorelix 78+78 | Cetrorelix 78+52 | Placebo
Number analyzed (Participants) | 211 | 226 | 213
Units on a scale | -4.0 (6.61) | -3.7 (5.90) | -3.8 (6.22)
Statistical Analysis 1: Comparison: Cetrorelix 78+78 vs Placebo; Test type: Superiority or Other; p = 0.7424, ANOVA; LS means estimate = -0.198, 95% CI 2-sided [-1.38 to 0.98]
Statistical Analysis 2: Comparison: Cetrorelix 78+52 vs Placebo; Test type: Superiority or Other; p = 0.926, ANOVA; LS means estimate = 0.055, 95% CI [-1.10 to 1.21]
Statistical Analysis 3: Comparison: Cetrorelix 78+78 vs Cetrorelix 78+52; Test type: Superiority or Other; p = 0.6699, ANOVA; LS means estimate = -0.252, 95% CI [-1.41 to 0.91]

2. Secondary Outcome: Time Course of Quality of Life
Description: The time course of quality of life: assessed by the following disease specific quality of life:"If you were to spend the rest of your life with the urinary conditions just the way it is now, how would you feel about that?" The rating scale is comprising a range of values from 0 to 6, with = delighted, 1 = pleased, 2 = mostly satisfied, 3 = mixed, 4 = mostly dissatisfied, 5 = unhappy, 6 = terrible.
Time Frame: Quality of life assessment in the following weeks: 4,12,26,30,38,46,52
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment Group A: Cetrorelix (CET) 78 mg + 78 mg: Treatment course 1: Cetrorelix 78 mg + 78 mg
  * Week 0: 52 mg CET (2 injections)
  * Week 2: 26 mg CET (1 injection)
  Treatment course 2:
  * Week 26: 52 mg CET (2 injections)
  * Week 28: 26 mg CET(1 injection)
    4 days with treatment, Day 1 of each indicated week, 6 injections in total per patient.
  Cetrorelix 78 mg + 78 mg
- Treatment Group B: CET 78 mg + 52 mg: Treatment course 1: Cetrorelix 78 mg + 52 mg
  * Week 0: 52 mg CET (2 injections)
  * Week 2: 26 mg CET (1 injection)
  Treatment course 2:
  * Week 26: 52 mg CET (2 injections)
  * Week 28: Placebo (1 injection)
    4 days with treatment, Day 1 of each indicated week, 6 injections in total per patient.
  Cetrorelix 78 mg + 52 mg
  Placebo
- Treatment Group C: Placebo: Treatment course 1:
  * Week 0: placebo (2 injections)
  * Week 2: placebo (1 injection)
  Treatment course 2:
  * Week 26: placebo (2 injections)
  * Week 28: placebo (1 injection)
    4 days with treatment, Day 1 of each indicated week, 6 injections in total per patient.
  Placebo
Arm/Group | Treatment Group A: Cetrorelix (CET) 78 mg + 78 mg | Treatment Group B: CET 78 mg + 52 mg | Treatment Group C: Placebo
Number analyzed (Participants) | 173 | 177 | 171
score on a scale
  Week 4 | -0.33 (1.16) | -0.42 (1.09) | -0.35 (1.00)
  Week 12 | -0.52 (1.21) | -0.67 (1.25) | -0.47 (1.05)
  Week 26 | -0.48 (1.18) | -0.70 (1.41) | -0.46 (1.07)
  Week 30 | -0.64 (1.20) | -0.71 (1.40) | -0.58 (1.24)
  Week 38 | -0.62 (1.20) | -0.77 (1.38) | -0.59 (1.22)
  Week 46 | -0.71 (1.28) | -0.67 (1.41) | -0.58 (1.20)
  Week 52 | -0.55 (1.25) | -0.62 (1.39) | -0.60 (1.11)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) related information will be collected during the entire course of the study. AEs will be reported as treatment-emergent adverse event (TEAE) if their start date ranges between the date of randomization and 3 months after the last administration of the study treatment. Adverse events (AEs) will be monitored from screening up to 90 weeks.
Description: For severity grading, the following definitions will be used:
  * Grade 1 - Mild: awareness of sign, symptom, or event, but easily tolerated
  * Grade 2 - Moderate: discomfort enough to cause interference usual activity and may warrant intervention
  * Grade 3 - Severe: incapacitating with inability to do usual activities or significantly affects clinical status and warrants intervention
  A special attention will be given to assess the severity of hot flashes.
Arm/Group | Cetrorelix 78+78 | Cetrorelix 78+52 | Placebo
Serious Adverse Events (participants affected / at risk) | 11/219 | 16/230 | 21/218
Other Adverse Events (participants affected / at risk) | 177/219 | 179/230 | 169/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetrorelix 78+78 (N=219) | Cetrorelix 78+52 (N=230) | Placebo (N=218)
IIIrd nerve paresis (Nervous system disorders) | 1 | 0 | 0
abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
angina pectoris (Cardiac disorders) | 0 | 2 | 0
asthenia (General disorders) | 0 | 0 | 1
asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
atrial flutter (Cardiac disorders) | 0 | 0 | 1
bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
blood bilirubin increased (Investigations) | 1 | 0 | 0
bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
cellulitis of legs (Infections and infestations) | 0 | 0 | 1
cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2
chest pain (General disorders) | 1 | 0 | 0
cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2
coronary artery disease (Cardiac disorders) | 1 | 4 | 0
decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 0 | 1
diverticulitis (Infections and infestations) | 0 | 0 | 1
gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
haematoma (Vascular disorders) | 1 | 0 | 0
hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
hypertensive emergency (Vascular disorders) | 0 | 1 | 0
hypotension (Vascular disorders) | 0 | 0 | 1
implant site infection (Infections and infestations) | 1 | 0 | 0
joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
mania (Psychiatric disorders) | 0 | 0 | 1
meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 1
muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1
myocardial infarction (Cardiac disorders) | 1 | 0 | 0
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
palpitations (Cardiac disorders) | 0 | 1 | 0
pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
pericarditis (Cardiac disorders) | 0 | 1 | 0
post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 2
prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
syncope (Nervous system disorders) | 1 | 0 | 0
transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2
urinary tract infection (Infections and infestations) | 0 | 1 | 0
urosepsis (Infections and infestations) | 0 | 0 | 1
vascular headache (Nervous system disorders) | 0 | 0 | 1
ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetrorelix 78+78 (N=219) | Cetrorelix 78+52 (N=230) | Placebo (N=218)
ALT increased (Investigations) | 1 | 5 | 1
Arthralgia (Skin and subcutaneous tissue disorders) | 11 | 8 | 10
Asthenia (General disorders) | 5 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 14 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 5
Diarrhea (Gastrointestinal disorders) | 12 | 15 | 6
Dizziness (Nervous system disorders) | 9 | 10 | 11
Erectile dysfunction (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 8
Fatigue (General disorders) | 5 | 5 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 6
Headache (Nervous system disorders) | 18 | 15 | 16
Hot flushes (Vascular disorders) | 9 | 10 | 6
Hypecholesterolemia (Metabolism and nutrition disorders) | 5 | 3 | 2
Hypertension (Vascular disorders) | 12 | 9 | 12
Inguinal hernia (Gastrointestinal disorders) | 2 | 1 | 5
Injection site pain (General disorders) | 21 | 17 | 8
Libido decreased (Psychiatric disorders) | 5 | 5 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 11 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 1
Nasopharyngitis (Infections and infestations) | 17 | 23 | 19
Nausea (Gastrointestinal disorders) | 4 | 5 | 9
Oedema peripheral (General disorders) | 5 | 4 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 7
PSA increased (Investigations) | 10 | 15 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5
Prostatitis (Reproductive system and breast disorders) | 5 | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 13 | 5 | 6
Sinusitis (Infections and infestations) | 3 | 12 | 2
Upper respiratory infection (Infections and infestations) | 16 | 15 | 13
Urinary retention (Renal and urinary disorders) | 6 | 3 | 2
Urinary tract infection (Infections and infestations) | 6 | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less